CLINICAL TRIAL: NCT04845334
Title: Complementary and Alternative Medicine Interventions in Targeting Pain
Acronym: CAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Scuola di Specializzazione in Psicologia Clinica dell'Università degli Studi di Torino (Unknown); Fondazione CRT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASO.Psg.15.01
Record Dates: First submitted 2021-02-03; First posted 2021-04-14 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Quadrantectomies; Spinal Fusion; Carotid Stenosis; Abdominal Aortic Aneurysm; Colectomy
Keywords: Relaxation response; Surgiva stress; Pain; Distress; Emotion regulation
MeSH Terms: conditions — Carotid Stenosis; Aortic Aneurysm, Abdominal; Pain; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical RR intervention (Experimental): Clinical RR intervention
  Interventions: Behavioral: RR intervention
- Standard care (No Intervention): Standard care

INTERVENTIONS:
Behavioral: RR intervention — The short psychological intervention consists of a narrative interview and a psychocorporeal intervention. Narrative interview: this is an interview aimed at exploring the experience and awareness of illness. The sharing of the dimension of pain and suffering, the verbalization of emotions, the narration of the history of illness, expectations and fears related to the intervention will be aimed at an emotional and cognitive restructuring of the experience of illness, improving the perception of internal resources and resilience.
  Psycho-corporeal intervention:it is a training to the psychophysiological technique of the "Relaxation Response" (R.R.) of Hebert Benson (Mind-Body Medical Institute of Havard), aimed at stress management and consequently at reducing the perception of pain
  Arms: Clinical RR intervention

SUMMARY:
This Controlled Randomized Clinical Trial aimed at determining the effectiveness of a modified RR intervention in reducing post-operative pain and psychological symptoms in patients undergoing surgery intervention.

Researches hypothesized that compared to controls patients undergoing modified RR intervention were characterized by

1. improved capability to discriminate emotions from bodily feelings;
2. reduce emotional distress;
3. reduced pain perception.

Moreover, researches hypothesized that (4) these effects were maintained over time.

DETAILED DESCRIPTION:
A Controlled Randomized Clinical Trial of a RR intervention for surgical patients was conducted in the SS. Antonio e Biagio e Cesare Arrigo Hospital, Alessandria, Italy.

Fifty-six patients were treated with the clinical RR intervention, while 62 patients were recruited as controls.

Variables were assessed through an ad hoc questionnaire and a pool of self-report questionnaires validated for the Italian population: the Toronto Alexithymia Scale (TAS-20), the Hospital Anxiety and Depression Scale (HADS), the Impact of Event Scale - Revised (IES-R), the Numeric Rating Scale (NRS), and the Emotion Thermometer (ET).

The TAS-20 is a frequently used 20-items self-report measure of alexithymia. A score ≥ 61 is considered to be indicative of alexithymia, whereas scores between 51 and 60 indicate borderline alexithymia. It has a 3-factor structure: Difficulty in Identifying Feelings (TAS-DIF); Difficulty in Describing Feelings (TAS-DDF), and Externally Oriented Thinking (TAS-EOT).

The HADS is a brief, reliable self-report measure used to assess anxiety and depression in hospitalized and ambulatory medical patients, as well as in primary care and research. It consists of 7 items for anxiety (HADS-A) and 7 for depression (HADS-D). Scores > 8 in each subscale are indicative of clinically relevant anxiety and depression, respectively.

The IES-R is a widely used 22-items self-report measure of subjective distress caused by traumatic events. It considers three independent dimensions: intrusion, avoidance, and hyper-arousal.

The NRS is a unidimensional measure of pain intensity in adults. It is a segmented numeric version of the visual analog scale (VAS), in which respondents select the number (0-10 integers) that best reflects the intensity of their pain. The common format is a horizontal bar or line.

The ET is a simple, self-report measure of four emotion domains (distress, anxiety, depression, and anger) and one non-emotion domain (need for help). Respondents have to rate each dimension on a vertical visual analogue scale (thermometer), with the anchors 0 and 10, to indicate which level of distress they experienced over the previous week.

Outcome measures were administered at 4 time-points:

T0: Baseline (3 months before the surgical intervention).

* Baseline alexithymia levels assessed with the TAS-20;
* baseline anxiety and depression levels assessed with the HADS;
* baseline post-traumatic distress assessed with the IES-R;
* baseline pain intensity assessed with the NRS;
* baseline psychological distress assessed with the ET;
* baseline use of analgesic drugs assessed with an ad hoc question.

T1: The morning before the surgical intervention.

* Changes in alexithymia levels assessed with the TAS-20;
* changes in anxiety and depression levels assessed with the HADS;
* changes in post-traumatic distress assessed with the IES-R;
* changes in pain intensity assessed with the NRS;
* changes in psychological distress assessed with the ET;
* changes in use of analgesic drugs assessed with an ad hoc question.

T2: At discharge, assessed up to 10 days.

* Changes in alexithymia levels assessed with the TAS-20;
* changes in anxiety and depression levels assessed with the HADS;
* changes in post-traumatic distress assessed with the IES-R;
* changes in pain intensity assessed with the NRS;
* changes in psychological distress assessed with the ET;
* changes in use of analgesic drugs assessed with an ad hoc question.

T3: 3 months after the surgical intervention.

* Changes in alexithymia levels assessed with the TAS-20;
* changes in anxiety and depression levels assessed with the HADS;
* changes in post-traumatic distress assessed with the IES-R;
* changes in pain intensity assessed with the NRS;
* changes in psychological distress assessed with the ET;
* changes in use of analgesic drugs assessed with an ad hoc question.

Subjects in the RR group underwent the clinical interventions between T0 and T1, while the controls underwent standard care.

Ethics

The study was reviewed and approved by the Institutional Review Board (IRB) of the SS. Antonio e Biagio e Cesare Arrigo Hospital, Alessandria, Italy. All participants gave informed written consent before entering the study. All research procedures were conducted in accordance with the ethical standards of the committees responsible for human experimentation (institutional and national) and with the Helsinki Declaration of 1975, as revised in 2008.

Participants

Patients were recruited between January 2015 and June 2017.

Patients in the Departments of Vascular Surgery, General Surgery and Neurosurgery were included, considering their similarities for what concerns surgical impact, recovery, and post-recovery expectation. Expected surgical patients in the recruitment period were computed considering the prevalent frequency of each specific intervention in every Department:

* General Surgery: patients scheduled for right hemicolectomies (60 patients/years expected), quadrantectomies (80 patients/years expected);
* Neurosurgery: patient scheduled for spinal fusion with non-traumatic etiology (225 patients/years expected)
* Vascular Surgery: patient scheduled for carotid stenosis or abdominal aortic aneurysm (205 patients/years expected).

With an expected population of 570 surgical patients in the recruitment period, an a priori power analysis conducted with G*Power (Faul et al., 2007) indicated that a total sample size of 82 participants was required (α = 0.05; 1-β = 0.80; d = 0.25).

Randomization and blinding:

A block randomization method was used with block size of 4, stratified by age, gender and clinical conditions. A series of numbers was generated in advance using a computer program. Following completion of the baseline measures, a research assistant assigned a study group to each participant, following the series generated by the computers. This research assistant as well as the personnel involved in the RR inspired intervention were aware of the patient-group assignment. Remaining study personnel were blind to subject's group assignment. In addition, for blinded purposes, the study participants were instructed not to discuss the intervention with anyone.

ELIGIBILITY:
Inclusion Criteria:

* patients waiting for a surgical intervention in the Departments of Vascular Surgery, General Surgery and Neurosurgery;
* age ≥ 18 years.

Exclusion Criteria:

* having a poor knowledge of the Italian language;
* having a cognitive impairment;
* having a certified psychiatric diagnosis;
* having a certified diagnosis of a neurodegenerative disease (i.e., Alzheimer disease, Parkinson disease, etc.)
* having been in psychiatric or psychological therapy in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in alexithymia (TAS scores) following a specific short psycho-corporeal intervention | Baseline; The morning before the surgical intervention; At discharge, assessed up to 10 days; 3 months after the surgical intervention
  Changes in the Toronto Alexithymia Scale (TAS-20) scores following a specific short psychocorporeal intervention
  * Total score. Range: 20-100. Higher scores mean a worse outcome.
  * Difficulty in Identifying Feelings (TAS-DIF). Range: 7-35. Higher scores mean a worse outcome.
  * Difficulty in Describing Feelings (TAS-DDF). Range: 5-25. Higher scores mean a worse outcome.
  * Externally Oriented Thinking (TAS-EOT). Range: 8-40. Higher scores mean a worse outcome.
Changes in anxiety and depression (HADS scores) following a specific short psycho-corporeal intervention | [Time Frame: Baseline; The morning before the surgical intervention; At discharge from the hospital, up to 10 days after the intervention; 3 months after the surgical intervention]
  Changes in the Hospital Anxiety and Depression Scale (HADS) scores following a specific short psycho-corporeal intervention.
  * Anxiety score. Range: 0-21. Higher scores mean a worse outcome.
  * Depression score. Range: 0-21. Higher scores mean a worse outcome.
Changes in post-traumatic distress (IES-R scores) following a specific short psycho-corporeal intervention | [Time Frame: Baseline; The morning before the surgical intervention; At discharge from the hospital, up to 10 days after the intervention; 3 months after the surgical intervention]
  Changes in the Impact of Event Scale - Revised (IES-R) scores following a specific short psycho-corporeal intervention
  * Total score. Range: 0-88. Higher scores mean a worse outcome.
  * Hyperarousal subscale. Range: 0-4. Higher scores mean a worse outcome.
  * Avoidance subscale. Range: 0-4. Higher scores mean a worse outcome.
  * Intrusion subscale. Range: 0-4. Higher scores mean a worse outcome.
Changes in pain intensity perception (NRS scores) following a specific short psycho-corporeal intervention | [Time Frame: Baseline; The morning before the surgical intervention; At discharge from the hospital, up to 10 days after the intervention; 3 months after the surgical intervention]
  Changes in the Numeric Rating Scale (NRS) scores following a specific short psycho-corporeal intervention
  • Total score. Range: 0-10. Higher scores mean a worse outcome.
Changes in psychological distress (ET scores) following a specific short psycho-corporeal intervention | [Time Frame: Baseline; The morning before the surgical intervention; At discharge from the hospital, up to 10 days after the intervention; 3 months after the surgical intervention]
  Changes in the Emotion Thermometer (ET) scores following a specific short psycho-corporeal intervention
  * Distress scale. Range: 0-10. Higher scores mean a worse outcome.
  * Anxiety scale. Range: 0-10. Higher scores mean a worse outcome.
  * Depression scale. Range: 0-10. Higher scores mean a worse outcome.
  * Anger scale. Range: 0-10. Higher scores mean a worse outcome.
  * Need for help scale. Range: 0-10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Effectiveness of the short psycho-corporeal intervention in reducing the use of analgesic drugs. | [Time Frame: Baseline; The morning before the surgical intervention; At discharge from the hospital, up to 10 days after the intervention; 3 months after the surgical intervention]
  Effectiveness of the short psycho-corporeal intervention in reducing the use of analgesic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Granieri, Professor, Study Director — Dipartimento di Psicologia dell'Università degli Studi di Torino; Fanny Guglielmucci, PhD, Study Director — Dipartimento di Psicologia dell'Università degli Studi di Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benson H, Beary JF, Carol MP. The relaxation response. Psychiatry. 1974 Feb;37(1):37-46. doi: 10.1080/00332747.1974.11023785. No abstract available. PMID 4810622
- [Background] Casey A, Chang BH, Huddleston J, Virani N, Benson H, Dusek JA. A model for integrating a mind/body approach to cardiac rehabilitation: outcomes and correlators. J Cardiopulm Rehabil Prev. 2009 Jul-Aug;29(4):230-8; quiz 239-40. doi: 10.1097/HCR.0b013e3181a33352. PMID 19451830
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Adamatti LC, Bandeira D, Ferreira MB. Preoperative predictors of moderate to intense acute postoperative pain in patients undergoing abdominal surgery. Acta Anaesthesiol Scand. 2002 Nov;46(10):1265-71. doi: 10.1034/j.1399-6576.2002.461015.x. PMID 12421200
- [Background] Chang BH, Casey A, Dusek JA, Benson H. Relaxation response and spirituality: Pathways to improve psychological outcomes in cardiac rehabilitation. J Psychosom Res. 2010 Aug;69(2):93-100. doi: 10.1016/j.jpsychores.2010.01.007. Epub 2010 Mar 1. PMID 20624507
- [Background] Glaros AG, Lumley MA. Alexithymia and pain in temporomandibular disorder. J Psychosom Res. 2005 Aug;59(2):85-8. doi: 10.1016/j.jpsychores.2005.05.007. PMID 16186003
- [Background] Honkalampi K, Hintikka J, Laukkanen E, Lehtonen J, Viinamaki H. Alexithymia and depression: a prospective study of patients with major depressive disorder. Psychosomatics. 2001 May-Jun;42(3):229-34. doi: 10.1176/appi.psy.42.3.229. PMID 11351111
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Lumley JW, Fielding GA, Rhodes M, Nathanson LK, Siu S, Stitz RW. Laparoscopic-assisted colorectal surgery. Lessons learned from 240 consecutive patients. Dis Colon Rectum. 1996 Feb;39(2):155-9. doi: 10.1007/BF02068069. PMID 8620781
- [Background] Tuzer V, Bulut SD, Bastug B, Kayalar G, Goka E, Bestepe E. Causal attributions and alexithymia in female patients with fibromyalgia or chronic low back pain. Nord J Psychiatry. 2011 Apr;65(2):138-44. doi: 10.3109/08039488.2010.522596. Epub 2010 Sep 27. PMID 20874000
- [Background] Villemure C, Bushnell CM. Cognitive modulation of pain: how do attention and emotion influence pain processing? Pain. 2002 Feb;95(3):195-199. doi: 10.1016/S0304-3959(02)00007-6. No abstract available. PMID 11839418
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Bagby RM, Taylor GJ, Parker JD. The Twenty-item Toronto Alexithymia Scale--II. Convergent, discriminant, and concurrent validity. J Psychosom Res. 1994 Jan;38(1):33-40. doi: 10.1016/0022-3999(94)90006-x. PMID 8126688
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Olsson I, Mykletun A, Dahl AA. The Hospital Anxiety and Depression Rating Scale: a cross-sectional study of psychometrics and case finding abilities in general practice. BMC Psychiatry. 2005 Dec 14;5:46. doi: 10.1186/1471-244X-5-46. PMID 16351733
- [Background] Craparo G, Faraci P, Rotondo G, Gori A. The Impact of Event Scale - Revised: psychometric properties of the Italian version in a sample of flood victims. Neuropsychiatr Dis Treat. 2013;9:1427-32. doi: 10.2147/NDT.S51793. Epub 2013 Sep 19. PMID 24092980
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Jensen MP, Moore MR, Bockow TB, Ehde DM, Engel JM. Psychosocial factors and adjustment to chronic pain in persons with physical disabilities: a systematic review. Arch Phys Med Rehabil. 2011 Jan;92(1):146-60. doi: 10.1016/j.apmr.2010.09.021. PMID 21187217
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Rodriguez CS. Pain measurement in the elderly: a review. Pain Manag Nurs. 2001 Jun;2(2):38-46. doi: 10.1053/jpmn.2001.23746. PMID 11706769
- [Background] Johnson C. Measuring Pain. Visual Analog Scale Versus Numeric Pain Scale: What is the Difference? J Chiropr Med. 2005 Winter;4(1):43-4. doi: 10.1016/S0899-3467(07)60112-8. PMID 19674646
- [Background] Mitchell AJ, Morgan JP, Petersen D, Fabbri S, Fayard C, Stoletniy L, Chiong J. Validation of simple visual-analogue thermometer screen for mood complications of cardiovascular disease: the Emotion Thermometers. J Affect Disord. 2012 Feb;136(3):1257-63. doi: 10.1016/j.jad.2011.06.008. Epub 2011 Jul 1. PMID 21723618
- [Background] Schubart JR, Mitchell AJ, Dietrich L, Gusani NJ. Accuracy of the Emotion Thermometers (ET) screening tool in patients undergoing surgery for upper gastrointestinal malignancies. J Psychosoc Oncol. 2015;33(1):1-14. doi: 10.1080/07347332.2014.977415. PMID 25396697
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343